CLINICAL TRIAL: NCT03933553
Title: Effect of Easy Sleep Complex Essential Oil Inhalation on Sleep Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kuang Tien General Hospital (Other)
Collaborators: Hung Kaung University (Other)
Responsible Party: Principal Investigator, Chun-pai Yang, MD, Head of Sleep Center, Kuang Tien General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: I10744
Record Dates: First submitted 2019-04-23; First posted 2019-05-01 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Sleep Disorder
Keywords: aromatherapy essential oil; Easy Sleep complex essential oil; Lavender essential oil; sleep disorders
MeSH Terms: conditions — Sleep Wake Disorders | interventions — Aromatherapy; Oils, Volatile

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Easy sleep complex essential oil (Experimental): Aromatherapy for 2 hours starting 10 minutes before sleep with 5 drops of the essential oil diluted in 50ml water
  Interventions: Other: Aromatherapy with essential oil
- Lavender essential oil (Active Comparator): Aromatherapy for 2 hours starting 10 minutes before sleep with 5 drops of the essential oil diluted in 50ml water
  Interventions: Other: Aromatherapy with essential oil

INTERVENTIONS:
Other: Aromatherapy with essential oil — the aromatherapy by fragrance inhalation

SUMMARY:
Sleep disorders affect human health tremendously. It has been reported that aromatherapy by fragrance inhalation can be used as an adjuvant therapy to modulate parasympathetic nervous activity for relieving stress and mood, and promoting sleep quality. Many researches confirmed that lavender essential oil can be used as an adjuvant therapy for sleep disorders. It can effectively relieve stress and modulate physical and mental status. However, many studies about aromatherapy lack sleep detection instruments to objectively confirm their effects on sleep physiology. Therefore, this study adopts Easy sleep complex essential oil as the experimental group. The lavender essential oil containing orange, petitgrain, rose, lavender, rosewood, ho wood, amyris essential oil and lavender oil is chosen as control group. The subjects will be randomly assigned to one of the two groups. The efficacy results will be evaluated and compared between the two groups. The investigators expect that aromatherapy by fragrance inhalation with Easy sleep complex essential oil will improve sleep quality more effectively than lavender essential oil.

DETAILED DESCRIPTION:
A Randomized, Single-blind, Active-Controlled Trial to Evaluate the aromatherapy by fragrance inhalation using Easy sleep complex essential oil in patients with sleep disorders.

ELIGIBILITY:
Inclusion Criteria:

* The subjects who signs the informed consent form approved by the Institutional Review Board.
* Adult between the ages of 20-65 with the ability to communicate and describe symptoms.
* The subjects has sleep disorders that last for at least three months and more than three nights per week.
* Pittsburgh Sleep Quality Index(PSQI) score greater than 5.
* The subjects are willing to cooperate with the study requirements, examinations and tests, including aromatherapy, polysomnography for two consecutive nights, questionnaire and blood tests.

Exclusion Criteria:

* The patients with abnormal olfactory system such as brain injury, acute or chronic sinusitis, and the history of nasal surgery.
* Patients who are currently taking sedatives or stimulant medicine or food such as coffee or refresh drink.
* Patients with a known history of allergy to aromatherapy or asthma.
* Patients has severe cardiovascular or pulmonary disease (e.g., cardiac failure or lung failure), or has cancer or other critical illness (e.g., renal dialysis).
* Pregnant or breastfeeding women.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2019-05-04 (Actual); Primary Completion 2022-01-17 (Actual); Study Completion 2022-01-17 (Actual)

PRIMARY OUTCOMES:
Electroencephalogram (EEG) | 2 days
  measure the alpha wave(8-14Hz), Vertex sharp wave(4-7Hz), K complex (negative- positive sharp component area), Spindle(7-14Hz for at least 0.5 sec), theta wave(4-7Hz), and delta wave(0.5-3Hz, amplitude>75uV).
Electrooculograph (EOG) | 2 days
  a record of the difference in electrical charge between the front and back of the eye
Electrocardiogram (ECG) | 2 days
  measure heart rate variability (HRV): change of R-R interval
Electromyogram (EMG) | 2 days
  recording the electrical activity produced by skeletal muscles
Respiratory effort | 2 days
  The amplitude change of chest and abdominal movement
Air flow | 2 days
  The amplitude change of nasal pressure and thermistor
Blood pressure (mmHg) | 2 days
  Systolic and Diastolic blood pressure
Blood oxygen saturation (the fraction of oxygen) | 2 days
  saturated hemoglobin relative to total hemoglobin in the blood
Heart Rate (beats per minute) | 2 days
  Rate of heart beat
The number of sleep gestures during the sleep | 2 days
  Analyzed with video recording overnight

SECONDARY OUTCOMES:
Concentration of Interleukin-1 | 2 days
  blood test with fasting status
Concentration of Interleukin-6 | 2 days
  blood test with fasting status
Concentration of Interleukin-8 | 2 days
  blood test with fasting status
Concentration of Tumor necrosis factor-alpha | 2 days
  blood test with fasting status
Concentration of Malonaldehyde | 2 days
  Indicator of oxidative stress
Concentration of Total antioxidant capacity | 2 days
  Indicator of oxidative stress

CONTACTS AND LOCATIONS:
Locations (1):
- Kuang Tien General Hospital, Taichung, Taiwan

REFERENCES:
- [Derived] Yang CP, Yang CC, Tsai IJ, Lin TH, Chiou YL, Wang HF, Chang CM, Yih KH. The immediate effects of lavender-based essential oil inhalation on subsequent polysomnography in people with poor sleep quality. J Chin Med Assoc. 2023 Jul 1;86(7):665-671. doi: 10.1097/JCMA.0000000000000932. Epub 2023 Apr 25. PMID 37098173